CLINICAL TRIAL: NCT02786069
Title: A Single-arm, Self-controlled, Three-period Dynamics Single-dose Escalation Safety and Pharmacokinetics Study for Propionyl L-carnitine Hydrochloride Tablets of Healthy Subjects in China
Brief Title: A Single-dose Escalation Safety and PK Study for PLC in Healthy Chinese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-201506-PLC-single dose
Record Dates: First submitted 2016-05-24; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Propionyl L-carnitine Hydrochloride

INTERVENTIONS:
Drug: Propionyl L-carnitine Hydrochloride — 500mg/ tablet; for oral administration, 1 dosage form is set for this trial: 1g, 2g and 4g.

SUMMARY:
The main objective is to evaluate the effect of single dose Propionyl-L-Carnitine Hydrochloride on clinical pharmacokinetic characteristics and its effect of clinical pharmacokinetic characteristics and safety on healthy Chinese subjects to provide a basis for market authorization registration.

DETAILED DESCRIPTION:
Before the official start of the study, to determine the appropriate dosing interval and a preliminary assessment of drug safety, first carried out the pre-trial, 4 subjects with different gender in half, after 7 days of run-in period, collect baseline background sampling point at day 4, no medication but water intake. At day 8 fasting oral propionyl L-carnitine hydrochloride tablets 0.5g, according to pre-designed schedule for blood samples, urine samples and clinical indicators, provide a reference for official trial.

Official trial is a single, open label, self-controlled, three-period, dose escalation, period fasting single oral administration trial. 12 chinese healthy adult subject met the inclusion criteria 12 people, each gender in half. Each subject first pass 7 days of run-in period, to eliminate the residual substances in food L-carnitine, stable baseline level of endogenous L-carnitine class substance within the subject; at day 4 was baseline sampling point, tno medication but water intake; at day 8 (1st period day 1) fasting oral propionyl L-carnitine hydrochloride tablets 1g; at day 12 (2nd period of day 1) fasting oral hydrochloride propionyl L-carnitine tablets 2g; the first 16 days (3rd period day 1) fasting oral propionyl L-carnitine hydrochloride tablets 4g.Throughout the trial period, control the subjects' diet, eating only allowed as far as possible food without substance L-carnitine class and drink boiled water,diet at sampling day 4, 8, 12, 16 need to be fixed consistently. Every 4 days of dosing interval washout period.

Subject need to follow blood, urine collection and diet control as required by protocol before the day of run-in period. During the trial should avoid vigorous exercise, meanwhile to avoid long-time bedding.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female, healthy subjects;
* Age: 19 to 45 years of age, of similar age;
* Weight: The weight of all subjects need ≥50 kg, body mass index [BMI = weight (kg) / height 2 (m 2)] within 19 to 24 kg / m2 range of weight as close as possible;
* Blood pressure: SBP 90-139mmHg, DBP 60-89 mmHg;
* The subjects must be informed consent before the trial, and voluntarily signed a written informed consent form;
* Subjects can be good communication with researchers and to complete the test in accordance with program requirements.

Exclusion Criteria:

Subjects having one or more cannot be selected for the trial:

Laboratory parameters:

* Before testing the safety evaluation of any one of the researchers baseline values considered clinically significant abnormalities;
* Hepatitis B surface antigen test positive;
* Hepatitis C antibody test positive;
* AIDS, syphilis testing positive;
* Pre-medication ECG abnormal situation at screening period or trial day 1 as followings:
* QTc> 450 ms (QTc using Bazett correction formula QTc = QT / RR0.5 computing);
* Ⅱ ° atrioventricular or Ⅲ ° atrioventricular block;
* heart rate <45 beats / min or> 100 beats / min;
* Room PR of> 200 ms or <110 ms;
* QRS complex> 120 ms;
* Pathological Q waves (in accordance with Q wave> 40 ms defined);
* Ventricular pre-excitation syndrome;

Medication history:

* 1 month before the trial orally used any inhibition or induction of hepatic drug metabolism of drugs;
* 2 weeks before the trial taking any medications (including prescription and non-prescription drugs and herbal preparations) persons;

Disease history and surgical history:

* Past history of suffering from structural heart disease, arrhythmias, heart failure, history of history, history of myocardial infarction, angina pectoris, history cannot be explained, fast ventricular reverse history, history of ventricular tachycardia, QT prolongation syndrome or have a history of long QT syndrome symptoms and family history (as evidenced by genetic or close relative at a young age due to cardiac causes of sudden death show);
* Have a history of thyroid disease or previously treated thyroid surgery;
* A history of immune system (such as a history of thymus disease);
* Within six months before the trial had received surgery;
* Have a history of severe digestive system diseases (such as having a significant clinical significance of gallbladder disease, known or suspected jaundice, hepatocellular adenoma, cavernous hemangioma of the liver and other liver diseases);
* Within six months before the trial have suffered from gastrointestinal or metabolic liver and kidney disease that can affect drug absorption (whether or not cured were excluded);
* Have any serious cardiovascular system, respiratory system, metabolic system and the nervous system a history;
* Suffering from blood coagulation disorders and other diseases system;
* Have a history of cancer;
* According to a clinical laboratory reference range limits, with hypokalemia, hypocalcemia;

Lifestyle:

* Within six months before the trial frequent drinkers, that drinking more than 14 units of alcohol a week (1 unit = 17.7 ml ethanol, or 1 unit = 357 ml alcohol content of 5% of the amount of alcohol in beer or 44 ml of 40% spirits or 147 ml alcohol content of 12% of the wine);
* Within three months before the trial daily cigarette consumption> one;
* Before the trial, 1 year history of drug abuse and drug taking too (such as marijuana, cocaine, opiates, benzodiazepines, amphetamines, barbiturates, tricyclic antidepressants, etc.);
* Before treatment 2 days to 8 days after drug overdose drinking tea, coffee and / or beverages containing caffeine (8 cups or more) every day;
* Eight days before treatment were drinking grapefruit juice and other beverages to medication after two days;

Others:

* Do not agree to take effective contraceptive measures after medication within 3 months;
* Allergies, including known allergies history to this drug excipients (microcrystalline cellulose, lactose, silica powder, sodium carboxymethyl starch, magnesium stearate);
* Within three months before the trial participated in any clinical trials or after the enrollment of this trial until 1 month after the end of the last follow-up visit to participate in other clinical trials;
* Before the trial within three months have donated blood, or planned to do so after until 1 month of the end of last follow-up visit;
* Have any food allergies or special dietary requirements, cannot comply with unified diets;
* The researchers judgments that those who should not be included;

Female subjects in addition to the above criteria, fulfilling any one of the following criteria must be excluded:

* Taking oral contraceptives before 1 month of trial;
* The use of long-acting estrogen or progestin injections or implants before 6 months of trial;
* Women of childbearing age failed to take adequate contraceptive measures before 2 weeks of trial;
* Women of childbearing age and their spouses do not agree to take following contraception measures within three months after medication: condoms, IUD;
* Pregnancy, lactation ;
* Urine pregnancy test was positive;

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | 0h, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24h after administration
  To observe area under curve characteristics of propionyl L-carnitine hydrochloride in single dose oral 1, 2, 4g

SECONDARY OUTCOMES:
cumulative excretion percentage | after drinking 0-2h, 2-4h, 4-8h, 8-12h, 12-24h for 4ml urine collection
  To estimate cumulative excretion percentage from the urine drug concentration in single dose oral 1, 2, 4g propionyl L-carnitine hydrochloride tablets

CONTACTS AND LOCATIONS:
Overall Officials: Heng-yan Qu, Principal Investigator — National Clinical Trial Institution of Affiliated Hospital of Military Medical Sciences